CLINICAL TRIAL: NCT03960996
Title: Long Term Effectiveness of Dacryocystorinostomy With and Without Bicanalicular Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-Dacryocystorinostomy; 22/RVO-FNOs/2019 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Lacrimal Duct Obstruction
Keywords: lacrimal duct obstruction; bicanalicular intubation; dacryocystorinostomy; silicone stent
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into two parallel groups.
Masking Description: No masking will be used in the course of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dacryocystorinostomy with bicanalicular intubation (Experimental): Patients with lacrimal duct obstruction enrolled into this study arm will undergo dacryocystorinostomy with bicanalicular intubation.
  Interventions: Procedure: dacryocystorinostomy
- Dacryocystorinostomy without bicanalicular intubation (Experimental): Patients with lacrimal duct obstruction enrolled into this study arm will undergo dacryocystorinostomy without bicanalicular intubation.
  Interventions: Procedure: dacryocystorinostomy

INTERVENTIONS:
Procedure: dacryocystorinostomy — Dacryocystorinostomy is a surgical procedure indicated in patients with lacrimal duct obstruction.

SUMMARY:
Dacryocystorinostomy (DCR) is an operation that is indicated for lacrimal duct obstruction. As a result of the lacrimal duct obstruction, tears are retained over the obstacle and repeated lacrimal infections occur. During DCR, the lacrimal sac is opened above the obliterated lacrimal duct and subsequently drained into the nasal cavity. The most common cause of unsuccessful surgery is intranasal stoma scarring. One of the methods that can increase the success rate of surgery is the introduction of silicone stent into the lacrimal duct during DCR, so-called bicanalicular intubation of the lacrimal system. The aim of the study is to compare long term effectiveness of DCR with and without bicanalicular intubation.

DETAILED DESCRIPTION:
Dacryocystorinostomy (DCR) is an operation that is indicated for lacrimal duct obstruction. Lacrimal duct obstruction can be caused by inflamation and trauma or might be the consequence of previous surgery in the lacrimal duct region. As a result of the lacrimal duct obstruction, tears are retained over the obstacle and repeated lacrimal infections occur. During DCR, the lacrimal sac is opened above the obliterated lacrimal duct and subsequently drained into the nasal cavity. The results of DCR are generally excellent and the success rate (regression of complaints) varies between 85-95% depending on the condition of the lacrimal pathways before surgery. Yet there is a constant effort to improve the results of operations. The most common cause of unsuccessful surgery is intranasal stoma scarring. It is caused by an inadequately formed bone window, an individual tendency to healing and scar formation, but a frequent cause is the insufficient opening of the tear bag or the formation of scars between the nasal septum and the lateral nasal wall. One of the methods that can increase the success rate of surgery is the introduction of silicone stent into the lacrimal duct during DCR, so-called bicanalicular intubation of the lacrimal system. Silicone stent remains in the lacrimal system for 12 weeks and prevents scarring. Results of previous studies are not clear whether bicanalicular intubation is beneficial. The aim of the study is to compare long term effectiveness of DCR with and without bicanalicular intubation.

ELIGIBILITY:
Inclusion Criteria:

* patients with lacrimal duct obstruction
* 18 to 79 years of age
* capable of general anesthesia
* signing of the informed consent

Exclusion Criteria:

- inability to undergo general anesthesia

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Recurrence of lacrimal duct obstruction at 6 months | 6 months
  The recurrence of lacrimal duct obstruction at 6 months after the procedure will be observed.
Recurrence of lacrimal duct obstruction at 12 months | 12 months
  The recurrence of lacrimal duct obstruction at 12 months after the procedure will be observed.
Recurrence of lacrimal duct obstruction at 24 months | 24 months
  The recurrence of lacrimal duct obstruction at 24 months after the procedure will be observed.
Recurrence of lacrimal duct obstruction at 36 months | 36 months
  The recurrence of lacrimal duct obstruction at 36 months after the procedure will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Komínek, prof.,MD,PhD,MBA, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Nomura K, Arakawa K, Sugawara M, Hidaka H, Suzuki J, Katori Y. Factors influencing endoscopic dacryocystorhinostomy outcome. Eur Arch Otorhinolaryngol. 2017 Jul;274(7):2773-2777. doi: 10.1007/s00405-017-4541-8. Epub 2017 Mar 20. PMID 28321534
- [Background] Coumou AD, Genders SW, Smid TM, Saeed P. Endoscopic dacryocystorhinostomy: long-term experience and outcomes. Acta Ophthalmol. 2017 Feb;95(1):74-78. doi: 10.1111/aos.13217. Epub 2016 Aug 29. PMID 27573690